CLINICAL TRIAL: NCT03508323
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase IV Study to Evaluate the Efficacy and Safety of Tenelia® in Patients Aged 65 and Older With Inadequately Controlled Type 2 Diabetes
Brief Title: Tenelia Elderly CGMS Study(TEDDY)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP_C403
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teneligliptin (Experimental)
  Interventions: Drug: Teneligliptin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teneligliptin — 20mg/qd
  Arms: Teneligliptin
Drug: Placebo — 1T/qd
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of Teneligliptin in Patients aged 65 and Older with inadequately controlled type 2 diabetes.

DETAILED DESCRIPTION:
To assess the efficacy and safety of Teneligliptin in Patients aged 65 and Older with inadequately controlled type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 65 years or older on screening
* Patients with type 2 diabetes mellitus
* Patients with 7.0% ≤ HbA1c ≤ 9.0% at the screening visit
* Patients with FPG < 270mg/dL on screening visit

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 12wks on baseline
  Change of HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: JH Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Bae JC, Kwak SH, Kim HJ, Kim SY, Hwang YC, Suh S, Hyun BJ, Cha JE, Won JC, Kim JH. Effects of Teneligliptin on HbA1c levels, Continuous Glucose Monitoring-Derived Time in Range and Glycemic Variability in Elderly Patients with T2DM (TEDDY Study). Diabetes Metab J. 2022 Jan;46(1):81-92. doi: 10.4093/dmj.2021.0016. Epub 2021 Jun 16. PMID 34130378